CLINICAL TRIAL: NCT03843528
Title: Epigenetic Modification for Relapse Prevention: a Dose-finding Study of Vorinostat Used in Combination With Low-dose Azacitidine in Children Undergoing Allogeneic Hematopoietic Cell Transplantation for Myeloid Malignancies
Brief Title: Vorinostat Dose-escalation After Allogeneic Hematopoietic Cell Transplantation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00202540
Record Dates: First submitted 2019-01-24; First posted 2019-02-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Mixed Phenotype Acute Leukemia; Juvenile Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Biphenotypic, Acute; Leukemia, Myelomonocytic, Juvenile | interventions — Vorinostat; Azacitidine

STUDY DESIGN:
Intervention Model Description: 3+3 dose-escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combined therapy (Experimental): Patients will be enrolled in blocks of 3, with vorinostat dose-escalation according to 3+3 study design.
  Low-dose azacitidine will be administered in a fixed dose to all patients, for days 1-5 of each 28 day cycle.
  Interventions: Drug: Vorinostat; Drug: Azacitidine Injection

INTERVENTIONS:
Drug: Vorinostat — Vorinostat will be administered concurrent with low-dose azacitidine post-transplant, on days 1-7 and 15-21 of 28 day cycles. This is an oral medication.
Drug: Azacitidine Injection — Azacitidine will be administered on days 1-5 of each 28 day cycle, either by IV or subcutaneous injection. The dose of azacitidine will be fixed, with no dose-escalation.

SUMMARY:
The objective of this study is to evaluate the maximum tolerated (MTD) of vorinostat used in combination with low-dose azacitidine after allogeneic hematopoietic cell transplantation (alloHCT) for prevention of relapse of childhood myeloid malignancies.

DETAILED DESCRIPTION:
Children and adolescents ages 1 to 21 years of age who are undergoing allogeneic hematopoietic cell transplantation for a myeloid malignancy (AML, MDS, JMML, MPAL) will be eligible. There are no restrictions on donor type, conditioning, stem cell source, of GVHD prophylaxis approach.

All participants will be treated on a single arm, and will initially receive 2 cycles of standard post-transplant azacitidine at a dose of 32mg/m2/dose IV/subcutnaeous for 5 days, in 28 day cycles. This is considered standard of care.

After tolerance of 2 cycles of azacitidine has been established, patients will be assigned to receive vorinostat orally at different dose levels, depending on the stage of the study. The dose level assignments will be conducted on a standard 3+3 design, whereby dose-escalation is peformed if previous patients tolerated the dose without dose-limiting toxicities, and dose-reduction is performed if dose-limiting toxicities are seen. The starting dose will be 100mg/m2/dose on days 1-7 and 15-21 of each 28 day cycles. This will be in addition to receiving azacitidine at the fixed dose above. In order to start each cycle, participants will be required to meet specific clinical parameters to ensure safety.

The dose of vorinostat between patients will be escalated or de-escalated until criteria for finding the maximum tolerated dose (MTD) is reached, and this will complete the study. Participants will continue to receive the prescribed dose of vorinostat for up to 7 cycles (9 total cycles of azacitidine).

Participants are followed for dose-limiting toxicities primarily during the first two course of combined therapy (cycles 3 and 4), but are continued to be tracked until the completion of all potential combined treatment (1 year or 7 combined cycles, whichever is earlier).

Principal aims:

1. To evaluate the maximum tolerated dose (MTD) of vorinostat used in combination with low-dose azacitidine after allogeneic hematopoietic cell transplantation (alloHCT) for childhood myeloid malignancies.

Secondary aims:

1. To describe the dose-limiting toxicities (DLT) of the vorinostat used in combination with low-dose azacitidine.
2. To describe rates of relapse, transplant related mortality, graft-versus-host disease, and overall survival.
3. To describe the effect of epigenetic modification on lymphocyte reconstitution in the post-alloHCT setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 1 year to 21 years of age.
2. Patient has a diagnosis of AML, MDS, MDS/AML, MPAL, or JMML. Note: patients are allowed to have received a HMA or HDACi prior to undergoing alloHCT.
3. Patient has undergone allogeneic hematopoietic cell transplantation (no restrictions on conditioning regimen, donor or stem cell source, or GVHD prophylaxis regimen).
4. Patient and/or parent(s) or legal guardian(s) are capable of understanding the study, including potential benefits and risks, and sign written informed consent. Age-appropriate assent will be obtained.
5. Female patient of childbearing potential has a negative screening pregnancy test (urine or serum, as per local institutional standard).
6. Female patient with infant(s) agrees not to breastfeed her infant(s) while on study.
7. Patient of child-bearing potential (male and female) agrees to use effective method of contraception during the study.

Exclusion Criteria:

1. Patient is enrolled on a clinical trial with investigational post-transplant medications. Note: trials involving defibrotide, post-transplant cyclophosphamide, and Lactobacillus plantarum are permitted. Other trials involving investigational medications that aren't leukemia or GVHD-directed may also be permitted after consultation with the overall PI.
2. Patient has a planned administration of non-protocol chemotherapy, radiation therapy, donor leukocyte infusion, or immunotherapy during the planned study period.
3. Patient has a known allergy to azacitidine or vorinostat.
4. Patient has chronic myelogenous leukemia.
5. Concomitant use of coumarin-derived anticoagulants or valproic acid.

   -

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 4 months
  The primary outcome of this study is to determine the MTD of vorinostat in combination with low-dose azacitidine, using dose-escalation methodology. This is based on toxicities developed by participants enrolled on the study.

SECONDARY OUTCOMES:
Dose-limiting toxicities | 4 months
  Rates of side effects from vorinostat will be recorded and described.
GVHD | 1 year
  Incidence of GVHD will be recorded and described.
Relapse | 1 year
  Incidence of relapse will be recorded and described
Survival | 1 year
  Duration of survival will be recorded and described
Immune recovery | 1 year
  Immune profile will be measured monthly for the first year post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Josephson, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No